CLINICAL TRIAL: NCT01419652
Title: Periprocedural Glycemic Control in Patients Undergoing Coronary Angiography With or Without Percutaneous Coronary Intervention
Brief Title: Periprocedural Glycemic Control in Patients Undergoing Coronary Angiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Steven Sedlis, Chief, Cardiology VA NYHHCS New York campus, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: bds1
Record Dates: First submitted 2011-08-12; First posted 2011-08-18 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes Mellitus; Coronary Artery Disease
Keywords: percutaneous coronary intervention
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- continue hypglycemic meds (Active Comparator)
  Interventions: Other: hold hypoglycemic meds
- control - hold drug (No Intervention)

INTERVENTIONS:
Other: hold hypoglycemic meds — continue versus hold hypoglycemic medications
  Arms: continue hypglycemic meds

SUMMARY:
There are 24 million people with diabetes mellitus (DM) in the United States. Over one-third of patients presenting for coronary angiography have known DM, and an additional 20% of patients without known DM present with hyperglycemia on the day of coronary angiography. Hyperglycemia in the setting of urgent and elective percutaneous coronary intervention (PCI) is associated with a 40% relative increase in long-term mortality regardless of diabetic status. Mechanisms linking periprocedural hyperglycemia to adverse outcomes are poorly understood and the effects of treatment are unknown. This is a pilot study aimed at determining the effectiveness, feasibility and safety of continuing long-acting hypoglycemic medications on the morning of coronary angiography. Since hyperglycemia may cause increased platelet reactivity, a secondary aim is to evaluate a possible mechanism of benefit of periprocedural glycemic control on platelet activity. Patients with DM on hypoglycemic medications undergoing coronary angiography will be randomized to either continue or hold their clinically-prescribed long-acting hypoglycemic medications on the day of procedure. Patients with and without DM will be randomized to either routine care or additional glycemic control with the Yale insulin infusion protocol for 6 hours post-PCI. The primary endpoint of this study will be mean blood glucose level at the time of arterial access in the hold versus continue groups. Secondary endpoints will be mean blood glucose level at 6 hours post-PCI in the Yale versus routine care groups and number of hypoglycemic events in the glycemic control versus no glycemic control groups. The exploratory analysis assessing the effect of glycemic control on platelet activity will guide further studies evaluating the translation of an individual's platelet phenotype to the clinical risk of increased long-term mortality following PCI. The outcomes for this study (glucose levels and platelet function) are all measured during the hospital stay which averages 1 day.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing coronary angiography at the Manhattan Campus of the VA NY Harbor Healthcare System

Exclusion Criteria:

* 1. Patients who do not or are unable to consent. 2. Patients participating in a competing study. 3. For platelet substudy, patients who took NSAIDs within 72 hours of blood collection or who are on cilostazol or dipyridamole as part of their routine medication regimen. 4. Patients with any other co-morbidities that would influence subject safety.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
periprocedural glucose | within 12 hours of randomization
  measure of blood glucose when cardiac catheterization begins at the time of arterial access

CONTACTS AND LOCATIONS:
Locations (1):
- VA New York Harbor, New York, New York, United States